CLINICAL TRIAL: NCT01162759
Title: Home Blood Pressure Monitoring Program
Brief Title: Home Blood Pressure Monitoring Project
Acronym: HBPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-08DMagi-01
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Hypertension
Keywords: hypertension, intervention
MeSH Terms: conditions — Hypertension | interventions — 4-(2-(4-hydroxybenzyl)-phenoxy)-N-methylbutylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): The control group receiving usual care
- Home Blood Pressure Monitoring Group (Experimental): Intervention group
  Interventions: Behavioral: Home Blood Pressure Monitoring

INTERVENTIONS:
Behavioral: Home Blood Pressure Monitoring — Home blood pressure readings are taken at least 3 times a week, uploaded to a Microsoft Health Vault account through American Heart Association Heart360 at least 1 time per week. Patients are followed by a clinical pharmacist, with physician oversight, who will make adjustments to antihypertensive medications or suggest additional medications using national JNC VII and KPCO hypertension guidelines.
  Other Names: HBPM
  Arms: Home Blood Pressure Monitoring Group

SUMMARY:
The goal of this project is to improve hypertension control at Kaiser Permanente Colorado (KPCO) by implementing a population-based multi-factorial intervention that uses home BP monitors that can download BP readings to KPCO's health records via internet, interactive voice response (IVR) technology, and multidisciplinary care team. Participants will be randomized to either the home blood pressure monitoring group receiving the multi-factorial intervention or the usual care group who will be receiving Kaiser standard of care. We will determine the proportion of patients in each group who achieve their target BP goals at 6 months, according to national clinical practice guidelines. The study hypothesis is that a higher proportion of patients with uncontrolled hypertension in the home blood pressure monitoring (HBPM) group will achieve their target blood pressure compared to those in the usual care (UC) group.

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

Primary:

• To determine the proportion of patients in each group who achieve their target BP goals at 6 months, according to national clinical practice guidelines

Secondary:

The following parameters will be evaluated between groups:

* Change in BP measures between baseline and at 6 months
* Proportion of patients who are receiving antihypertensive treatments in accordance to national clinical practice guidelines
* Adherence to hypertensive medication regimen during the 6-month follow-up period
* Patient satisfaction with the care model.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years At least 1 diagnosis for hypertension,

  * Receive primary care from one of the participating clinics,
  * The two most recent BPs documented within that last 24 months are elevated (SBP>140 and/or DBP>90)
  * Receiving < 3 antihypertensive medications, and
  * Have access to a computer with a USB port.

Exclusion Criteria:

* Pregnant, or breast-feeding,
* Patients on dialysis or being followed by nephrology,
* Patients with coronary artery disease, given these patients are already followed by the Clinical Pharmacy Cardiac Risk Service (CPCRS),
* On KPCO "Do Not Call" or deceased list,
* PCP does not give permission to include patient in the study,
* BP is at or below target at the baseline study visit,
* Not English-speaking.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
BP at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David J Magid, MD, MPH, Principal Investigator — Kaiser Permanente; Kari Olson, PharmD, Principal Investigator — Kaiser Permanente; Sarah J Billups, PharmD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Colorado, Institute of Health Research, Denver, Colorado, United States

REFERENCES:
- [Derived] Magid DJ, Olson KL, Billups SJ, Wagner NM, Lyons EE, Kroner BA. A pharmacist-led, American Heart Association Heart360 Web-enabled home blood pressure monitoring program. Circ Cardiovasc Qual Outcomes. 2013 Mar 1;6(2):157-63. doi: 10.1161/CIRCOUTCOMES.112.968172. Epub 2013 Mar 5. PMID 23463811